CLINICAL TRIAL: NCT07371364
Title: Development and Evaluation of the Effectiveness of a Health Promotion Model Based Mobile Application for Women With Polycystic Ovary Syndrome
Brief Title: Mobile Application for Women With Polycystic Ovary Syndrome
Acronym: Polycystic
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, merve yilmaz menek, Assoc. Prof., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-1425; 224S421 (Other Grant/Funding Number: TUBITAK 1002-A)
Record Dates: First submitted 2026-01-12; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Women Health; Polycystic Ovary Syndrome (PCOS); Physiotherapy and Rehabilitation; Dietetics; Mobile Application
Keywords: Polycystic Ovary Syndrome; Mobile application; Exercises; nutrition; health promotion
MeSH Terms: conditions — Polycystic Ovary Syndrome; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Mobile application (Experimental): Women with PCOS in this group will be included in a regular exercise and nutrition program for 8 weeks using the mobile application.
  The development and use of the mobile application by women with PCOS consists of several components:
  1. Preparation and development of the mobile application content
  2. Health coaching within the mobile application
  3. Creation of exercise content within the mobile application
  4. Creation of a nutrition program within the mobile application
  5. Completion of evaluation forms via the mobile application
  6. Obtaining reports on participants via the mobile application
  Interventions: Other: Mobile application
- Group 2: Control group (Experimental): The control group will be given a PCOS-specific exercise or nutrition program booklet.
  Interventions: Other: control group

INTERVENTIONS:
Other: Mobile application — Women with PCOS in this group will be included in a regular aerobic and strengthening exercises and nutrition program for 8 weeks using the mobile application.
  Arms: Group 1: Mobile application
Other: control group — The control group will be given a PCOS-specific exercises or nutrition program via a handout.
  Arms: Group 2: Control group

SUMMARY:
Objective: The aim is to develop a mobile application based on the Health Promotion Model for the management of PCOS and to determine the effect of this application on improving nutrition and exercise behavior in women with PCOS.

Method: The study population will consist of 114 women diagnosed with PCOS according to the Rotterdam criteria (2003) by a specialist in Obstetrics and Gynecology (G power 3.1.9.7). Inclusion criteria are being over 18 years old, female, diagnosed with PCOS, willingness to participate in the study, owning a smartphone with Android or iOS operating system, having digital literacy, and not having a diagnosed psychiatric condition. Exclusion criteria include being pregnant or planning to become pregnant during the study, having musculoskeletal, neurological, respiratory, or cardiovascular diseases, undergoing any surgery or having health issues that could affect physical activity for more than a month, unwillingness to participate in the study for any reason, and not having internet access. Participants will be randomly assigned to either the experimental or control group. The experimental group will receive a PCOS-specific exercise and nutrition program through the mobile app based on the Health Promotion Model, while the control group will receive the program via a pamphlet and it will be applied over 8 weeks. The mobile application will include an exercise program, nutrition counseling, and health coaching for PCOS management, all aligned with the Health Promotion Model. At the beginning and end of the study, participants' blood measurements, anthropometric measurements, physical activity levels, exercise behavior, and adherence to the Mediterranean Diet will be evaluated.

DETAILED DESCRIPTION:
Introduction: Polycystic ovary syndrome (PCOS) is a lifelong endocrine disorder affecting 10 to 15% of women worldwide. Women with PCOS experience a range of physical and psychological issues, including hirsutism, acne, menstrual irregularities, hair loss, insulin resistance, metabolic syndrome, cardiovascular diseases, obesity, bipolar disorder, anxiety, depression, as well as sexual dysfunction and decreased quality of life. The most common problems associated with PCOS are menstrual irregularities, infertility, obesity, type 2 diabetes mellitus (T2DM), and metabolic syndrome. The primary goal of PCOS management is to improve hormonal and metabolic status, prevent future comorbid complications, and enhance the quality of life for young women with PCOS (Meczekalski et al. 2023). Literature review indicates that one of the most effective ways to improve quality of life in patients is through model-based educational interventions. In this context, one of the most comprehensive and widely used models for patient education provided by nurses is Pender's "Health Promotion Model." By creating a mobile application that facilitates adherence to physical activity and diet programs in the management of PCOS, it is expected to alleviate PCOS symptoms and improve women's quality of life.

Objective: The aim is to develop a mobile application based on the Health Promotion Model for the management of PCOS and to determine the effect of this application on improving nutrition and exercise behavior in women with PCOS.

Method: The study population will consist of 114 women diagnosed with PCOS according to the Rotterdam criteria (2003) by a specialist in Obstetrics and Gynecology (G power 3.1.9.7). Inclusion criteria are being over 18 years old, female, diagnosed with PCOS, willingness to participate in the study, owning a smartphone with Android or iOS operating system, having digital literacy, and not having a diagnosed psychiatric condition. Exclusion criteria include being pregnant or planning to become pregnant during the study, having musculoskeletal, neurological, respiratory, or cardiovascular diseases, undergoing any surgery or having health issues that could affect physical activity for more than a month, unwillingness to participate in the study for any reason, and not having internet access. Participants will be randomly assigned to either the experimental or control group. The experimental group will receive a PCOS-specific exercise and nutrition program through the mobile app based on the Health Promotion Model, while the control group will receive the program via a pamphlet and it will be applied over 8 weeks. The mobile application will include an exercise program, nutrition counseling, and health coaching for PCOS management, all aligned with the Health Promotion Model. At the beginning and end of the study, participants' blood measurements, anthropometric measurements, physical activity levels, exercise behavior, and adherence to the Mediterranean Diet will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being over 8 years old,
* Being female,
* Having a PCOS diagnosis,
* Volunteering to participate in the study,
* Having a mobile phone with Android or iOS operating system,
* Having computer literacy (good phone usage skills),
* Not having a diagnosed psychiatric illness.

Exclusion Criteria:

* Pregnancy or planning to become pregnant during the study period,
* The participant having a musculoskeletal, neurological, respiratory, or cardiovascular disease,
* Having any surgery or health problem that would affect their ability to be physically active for more than one month, The participant not wanting to participate in the study for any reason,
* The participant not having internet access.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility is based on biological sex due to the pathophysiology of PCOS.
Enrollment: 92 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) assesment | From enrollment to the end of treatment at 8 weeks
  Participants' BMI will be calculated by dividing body weight (kg) by the square of their height in meters. It will be reported as kg/m^2)
Waist circumference measurement | From enrollment to the end of treatment at 8 weeks
  Waist circumference measurement will be performed with a measuring tape while the participant is standing. The measurement will be taken by locating the lowest rib cage on the right side of the body and the iliac crest and determining the midpoint between these points. It will be reported as cantimeter.
Hip circumference measurement | From enrollment to the end of treatment at 8 weeks
  Hip circumference measurement will be taken with a measuring tape while the person is standing on their side, at the widest part of their hips. It will be reported as cantimeter.
The International Physical Activity Questionnaire | From enrollment to the end of treatment at 8 weeks
  It which measures physical activity level, consists of 4 separate sections and a total of 7 questions. It assesses how many days in the past week, and for how long each day, individuals engaged in vigorous physical activity (PPE), moderate-intensity physical activity (MOI), and walking (W). The final question determines the time spent without movement (sitting, lying down, etc.). MET (Metabolic Equivalent Minutes) is used to determine physical activity level. 1 MET = 3.5 ml/kg/min. By determining how many days a week and for how long individuals engaged in vigorous physical activity, moderate-intensity physical activity, and walking, the total amount of METs expended from these three different physical activities is calculated. Physical activity level is determined in 3 categories: Category 1: Inactive (<300 MET-min/week), Category 2: Minimally Active (600-3000 MET-min/week), and Category 3: Always Active (>3000 MET-min/week).
Exercise Behavior Assessment | From enrollment to the end of treatment at 8 weeks
  This will be assessed using the Exercise Behavior Change Stages Questionnaire. This questionnaire was developed by Marcus and Lewis to identify the stages of exercise behavior (Marcus and Lewis, 2003). The questionnaire consists of four items. The items, which aim to determine participants' willingness to exercise, are answered with yes/no. Individuals are divided into five separate exercise behavior stages based on their responses to the items, according to their intentions and habits regarding exercise: Pre-tendency, Tendency, Preparation, Movement, and Continuity. The questions asked in the questionnaire are as follows: 1. I am currently engaged in moderate physical activity. 2. I intend to increase my participation in moderate physical activity within 6 months. 3. I am currently regularly engaged in moderate physical activity. 4. I have been regularly engaged in moderate physical activity for the last 6 months.
Adherence to the Mediterranean Diet | From enrollment to the end of treatment at 8 weeks
  Participants' adherence to the Mediterranean diet will be assessed using the 14-item Mediterranean Diet Adherence Scale (MEDAS), developed by Martínez-González et al. for the PREDIMED study. The 14 questions on the scale will be administered by the researcher through face-to-face interviews with individuals. The Mediterranean Diet Adherence Scale scoring range is 0-14 points. Diet adherence scores of <5 will be considered poor adherence, 6-9 moderate adherence, and ≥10 good adherence.
Blood measurements | From enrollment to the end of treatment at 8 weeks
  Assessment of insulin resistance and lipid profile; Fasting glucose, Glycated Hemoglobin (HbA1c), HOMA-IR will be done.

CONTACTS AND LOCATIONS:
Overall Officials: MERVE YILMAZ MENEK, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will not share the individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Lee H, Lee SH. Effectiveness of an Integrated Mobile Application for Lifestyle Modifications in Overweight Women with Polycystic Ovarian Syndrome: A Randomized Controlled Trial. Life (Basel). 2023 Jul 10;13(7):1533. doi: 10.3390/life13071533. PMID 37511908
- See also: Effectiveness of an Integrated Mobile Application for Lifestyle Modifications in Overweight Women with Polycystic Ovarian Syndrome: A Randomized Controlled Trial — http://pubmed.ncbi.nlm.nih.gov/37511908/
- Available data/document: Study Protocol — http://pubmed.ncbi.nlm.nih.gov/37511908/ — IPD data may be provided by the principal investigator if required.